CLINICAL TRIAL: NCT07108296
Title: Multi-center Clinical Cohort Study on Cardiopulmonary Exercise Tolerance Standards in Chinese Healthy Population
Brief Title: A Study on Cardiopulmonary Exercise Tolerance Standards for Healthy Chinese Population
Acronym: MCCS-CCPETS
Status: Not yet recruiting | Type: Observational
Sponsor: Affiliated Hospital of Changchun University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoping Meng, Head of Cardiac Rehabilitation Department, Affiliated Hospital of Changchun University of Chinese Medicine
Other Study IDs: KFKT-2025-KY-010; KFKT-2025-KY-010 (Other Grant/Funding Number: China Rehabilitation Medicine Association)
Record Dates: First submitted 2025-08-04; First posted 2025-08-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Oxygen Consumption; Cardiorespiratory Fitness
Keywords: Peak Oxygen Uptake; VO2@AT; Cardiopulmonary Exercise Tolerance; Prediction Model; Healthy Population
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese Age-Sex-Stratified Cardiopulmonary Function Cohort (CACSF Cohort)
  Interventions: Other: cardiopulmonary exercise testing (CPET)

INTERVENTIONS:
Other: cardiopulmonary exercise testing (CPET) — In this study, the cardiopulmonary exercise testing (CPET) system used breath-by-breath continuous analysis for gas exchange and ventilation variables. The protocol included spirometry with an 8-breath data collection method. The cycle ergometer workload ranged from 10 to 40 W/min using a RAMP protocol. The standard CPET protocol comprised a 3-min rest, 3-min warm-up, 8 - 12 min incremental exercise phase, and 3-min each of active and passive recovery.

SUMMARY:
This project intends to conduct a large-sample, prospective, multicenter clinical cohort study in healthy populations. By utilizing a digital cardiopulmonary rehabilitation clinical data research platform, The investigators aim to achieve automated, standardized, and uniform collection, analysis, and AI modeling of large-scale cardiopulmonary exercise testing (CPET) data. The ultimate goals are:

To establish reference standards for cardiopulmonary exercise capacity in the Chinese healthy population.

To develop machine learning-based predictive models for key CPET variables (e.g., peak VO₂) tailored to Chinese demographics.

To compare performance differences between domestically produced and imported CPET devices.

ELIGIBILITY:
Inclusion Criteria:

* Detailed medical history taken, with no symptoms of discomfort reported
* Good physical condition, with no history of severe chronic diseases
* No history of long - term medication use
* Willing to undergo cardiopulmonary exercise testing, with no ST - T segment changes observed during the test
* Age: 18 - 65 years old
* BMI: 18.5 - 28kg/m²
* No smoking history or quit smoking for ≥5 years
* Physical examination reports within 2 years show no significant abnormalities.

Exclusion Criteria:

* Pre - test resting blood pressure ≥160/100 mmHg (1 mmHg=0.133 kPa)
* Chronic cardiovascular diseases, such as heart failure, coronary atherosclerotic heart disease, hypertension, congenital heart disease, cardiomyopathy, and severe arrhythmias
* Respiratory diseases, such as chronic obstructive pulmonary disease, asthma, pulmonary artery hypertension, bronchiectasis, and respiratory failure
* Digestive system diseases, such as peptic ulcer, gastrointestinal bleeding, hepatitis, liver cirrhosis, ulcerative colitis, Crohn's disease, chronic pancreatitis, and chronic cholecystitis
* Endocrine system diseases, such as hyperthyroidism, hypothyroidism, diabetes, and other diseases with clear hormone abnormalities
* Acute or chronic kidney diseases, blood system diseases, malignant tumors, and bone and joint diseases that affect activity
* No history of acute infection within 2 weeks
* Unable to cooperate with the examination
* Contraindications to cardiopulmonary exercise testing: acute myocardial infarction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals aged 18 - 65.
Sampling Method: Probability Sample
Enrollment: 4620 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen Uptake | On the day of enrollment
  When measuring the peak oxygen uptake of healthy people with a cycle ergometer, first ensure participants are healthy and have signed consent forms. Prepare the cycle ergometer and other equipment, adjusting them to a suitable position. After a 3 - minute warm - up, start the incremental loading test, which lasts 8 - 12 minutes, until termination criteria are met. Record the data, calculate the peak oxygen uptake, and assess the cardiopulmonary function.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Quanzhou First Hospital Affiliated to Fujian Medical University, Quanzhou, Fujian
  - Guangdong Provincial People's Hospital Affiliated to Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Jiangbin Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The Second Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Anyang Regional Hospital of Puyang City, Henan Province, Puyang, Henan
  - Zhengzhou Central Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Second Hospital of Central South University, Changsha, Hunan
  - Affiliated Hospital of Changchun University of Chinese Medicine, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shangdong
  - Tongji Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No
all IPD collected throughout the trial, only IPD used in the results publication

REFERENCES:
- [Background] Strain T, Flaxman S, Guthold R, Semenova E, Cowan M, Riley LM, Bull FC, Stevens GA; Country Data Author Group. National, regional, and global trends in insufficient physical activity among adults from 2000 to 2022: a pooled analysis of 507 population-based surveys with 5.7 million participants. Lancet Glob Health. 2024 Aug;12(8):e1232-e1243. doi: 10.1016/S2214-109X(24)00150-5. Epub 2024 Jun 25. PMID 38942042
- [Background] Weeldreyer NR, De Guzman JC, Paterson C, Allen JD, Gaesser GA, Angadi SS. Cardiorespiratory fitness, body mass index and mortality: a systematic review and meta-analysis. Br J Sports Med. 2025 Feb 20;59(5):339-346. doi: 10.1136/bjsports-2024-108748. PMID 39537313
- [Background] Wang J, Ren C, Xu S, Yuan Y, Song Y, Xie D, Wang K, Yuan L, Shen T, Xu L, Tang Y, Gao W, Zhao W. A reference equation for peak oxygen uptake for cycle ergometry in Chinese adult participants. Sci Rep. 2025 Mar 29;15(1):10876. doi: 10.1038/s41598-025-94207-7. PMID 40157952
- [Background] Brazile TL, Levine BD, Shafer KM. Cardiopulmonary Exercise Testing. NEJM Evid. 2025 Feb;4(2):EVIDra2400390. doi: 10.1056/EVIDra2400390. Epub 2025 Jan 28. PMID 39873542
- [Background] Kokkinos P, Kaminsky LA, Arena R, Zhang J, Myers J. A new generalized cycle ergometry equation for predicting maximal oxygen uptake: The Fitness Registry and the Importance of Exercise National Database (FRIEND). Eur J Prev Cardiol. 2018 Jul;25(10):1077-1082. doi: 10.1177/2047487318772667. Epub 2018 Apr 25. PMID 29692203
- [Background] Kaminsky LA, Myers J, Arena R. Determining Cardiorespiratory Fitness With Precision: Compendium of Findings From the FRIEND Registry. Prog Cardiovasc Dis. 2019 Jan-Feb;62(1):76-82. doi: 10.1016/j.pcad.2018.10.003. Epub 2018 Oct 30. PMID 30385268
- [Background] Daneshvar F, Weinreich M, Daneshvar D, Sperling M, Salmane C, Yacoub H, Gabriels J, McGinn T, Smith MC. Cardiorespiratory Fitness in Internal Medicine Residents: Are Future Physicians Becoming Deconditioned? J Grad Med Educ. 2017 Feb;9(1):97-101. doi: 10.4300/JGME-D-15-00720.1. PMID 28261402
- [Background] de Souza E Silva CG, Kaminsky LA, Arena R, Christle JW, Araujo CGS, Lima RM, Ashley EA, Myers J. A reference equation for maximal aerobic power for treadmill and cycle ergometer exercise testing: Analysis from the FRIEND registry. Eur J Prev Cardiol. 2018 May;25(7):742-750. doi: 10.1177/2047487318763958. Epub 2018 Mar 8. PMID 29517365
- [Background] Ashikaga K, Itoh H, Maeda T, Itoh H, Ichikawa Y, Tanaka S, Ajisaka R, Koike A, Makita S, Omiya K, Kato Y, Adachi H, Nagayama M, Tajima A, Harada N, Akashi YJ; Committee on Exercise Prescription for Patients (CEPP) Members. Ventilatory efficiency during ramp exercise in relation to age and sex in a healthy Japanese population. J Cardiol. 2021 Jan;77(1):57-64. doi: 10.1016/j.jjcc.2020.07.008. Epub 2020 Aug 5. PMID 32768174
- [Background] Katzmarzyk PT, Friedenreich C, Shiroma EJ, Lee IM. Physical inactivity and non-communicable disease burden in low-income, middle-income and high-income countries. Br J Sports Med. 2022 Jan;56(2):101-106. doi: 10.1136/bjsports-2020-103640. Epub 2021 Mar 29. PMID 33782046